CLINICAL TRIAL: NCT01678339
Title: Sicilian Administrative Data Base Study in Acute Coronary Syndrome Patients
Acronym: HEALTH-DB ACS
Status: Withdrawn | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CIT-XXX-2012/1
Record Dates: First submitted 2012-08-23; First posted 2012-09-05 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Acute Coronary Syndrome; Acute Myocardial Infarction
Keywords: ACS; AMI
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
Thi is an observational, non interventional, cohort analysis by using administrative databases (drugs treatment, laboratory and diagnostic tests, specialist visits and hospitalizations) of Sicilia region to evaluate treatment patterns of patients after Acute Coronary Syndrome (ACS) event.

DETAILED DESCRIPTION:
HEALTH-DB ACS

ELIGIBILITY:
Inclusion Criteria:

* Subjects discharged alive from hospitalization for ACS

Exclusion Criteria:

* All patients that don't have a continuative presence as beneficiaries of the region between January 1st, 2007 and December 31st 2011 will be excluded from analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients discharged alive from an hospitalization for Acute Myocardial Infarction (AMI) between January, 1st 2008 and December, 31st 2010 (inclusion period) will be included into analysis. The discharge date will be defined as "inclusion date".
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-09; Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
The diagnostic path for each patient included in the analysis will be described by using all prescription for laboratory test (eg. total cholesterol, LDL cholesterol) and/or diagnostics tests (eg. electrocardiogram) during the observation period. | up to 2 years
The drugs treatment path will be described by using all prescriptions of antihypertensive drugs, lipid-lowering drugs and antiplatelet drugs during the observation period. | up to 2 years
Adherence to treatment will be calculated in the manner suggested by the literature and used in previous publications. Different methods of assessment will, however, used in order to study the variability of results. The analysis will be conducted over | up to 2 years
The chronological analysis of the requirements will allow the identification of potential therapeutic combinations or substitutions. | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Flore La Tour, Study Chair — AstraZeneca CLINICAL RESEARCH DIRECTOR; Raffaele Sabia, Study Director — AstraZeneca Italy - VP MEDICAL; Rosalia Traiana, Doctor of Pharmacology, Principal Investigator — Department of Pharmaceutical Health - SICILIAN REGION
Locations (1):
- Research Site, Palermo, Italy